CLINICAL TRIAL: NCT05486702
Title: The Effects of Different Time-Restricted Eating Schedules With Exercise on the Body Composition in Overweight Adults
Brief Title: Time-Restricted Eating With Exercise
Acronym: TRE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Georgia College and State University (Other)
Responsible Party: Principal Investigator, Jinkyung Park, Assistant Professor, Georgia College and State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FRG202132
Record Dates: First submitted 2022-06-22; First posted 2022-08-03 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Time Restricted Eating (Experimental): 8-hour eating period from 7 am to 3 pm with exercise
  Interventions: Other: Time Restricted Eating
- Late Time Restricted Eating (Experimental): 8-hour eating period from 3 pm to 11 pm with exercise
  Interventions: Other: Time Restricted Eating

INTERVENTIONS:
Other: Time Restricted Eating — Time restricted eating (TRE) can be divided into early TRE (eTRE) and late TRE (lTRE), depending on the time of day of the eating window.

SUMMARY:
The purpose of the study is to determine if body composition differs between early time restricted eating (8-hour feeding period from 7 am to 3 pm) with exercise and late time restricted eating (8-hour feeding period from 3 pm to 11 pm) with exercise in overweight adults.

DETAILED DESCRIPTION:
Time-restricted eating (TRE) is a hot trend in weight-loss diets. TRE can reduce cardio-metabolic risks, thereby lowering body weight, blood pressure, lipid profile, glucose, and inflammation. The most effective way for the overweight population to improve body composition is to incorporate TRE with exercise. However, there were only two TRE interventions in humans that included exercise, suggesting that the additive effect of TRE to exercise may be dependent on dietary timing. TRE can be divided into early TRE (eTRE) and late TRE (lTRE), depending on the time of day of the eating window. However, whether different TRE schedules with exercise can improve cardio-metabolic health is questionable. There have been no interventions of different TRE schedules with exercise. This study will be beneficial for determining which TRE schedule with exercise is efficacious to prevent cardio-metabolic disease.

ELIGIBILITY:
Lists of inclusion criteria: the participants will be allowed to participate in this study if they

1. are adults, aged between 18-30 years
2. are apparently healthy and physically inactive (defined as any form of physical activity performed < 2 days per week)
3. are overweight (BMI 25-<30 kg/m2)
4. are non-smokers
5. are free from the following chronic medical conditions: heart disease, arrhythmias, diabetes, thyroid disease, bleeding disorder, history of pulmonary disease, hypertension, hepatorenal disease, musculoskeletal disorder, neuromuscular/neurological disease, autoimmune disease, cancer, peptic ulcers, anemia, or chronic infection (HIV)
6. are free from the orthopedic conditions that would hinder physical activity
7. have not taken any heart, pulmonary, thyroid, anti-hyperlipidemic, hypoglycemic, anti-hypertensive, endocrinological (e.g, thyroid, insulin, etc), emotional/psychotropic (e.g,Prednisone, Ritalin, Adderall), neuromuscular/neurological, or androgenic medications(anabolic steroids)
8. have low risk for cardiovascular disease and with no contraindications to exercise as outlined by the American College of Sports Medicine (ACSM) will be included.

Lists of exclusion criteria: the participants will not be allowed to participate in this study if they

1. are younger than 18 years and older than 30 years.
2. have consumed any medication for chronic medical condition.
3. are participating in weight management programs.
4. have constrictions to exercise.
5. are currently exercising regularly (at least 2 days per week).

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-08 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in body composition on the dual-energy X-ray absorptiometry (DXA) at week 10 | Baseline and Week 10
  The DXA is a validated instrument, assessing fat, soft tissue, and bone mass.

CONTACTS AND LOCATIONS:
Overall Officials: Jinkyung Park, Dr., Principal Investigator — Georgia College and State University
Locations (3):
- United States (3):
  - Exercise Science Laboratory, Milledgeville, Georgia
  - Clinical Research Laboratory, Syracuse, New York
  - Anatomical Laboratory, Wichita Falls, Texas

IPD SHARING:
Plan to Share IPD: No